CLINICAL TRIAL: NCT05832879
Title: A Pilot Study of Telehealth Treatment for Opioid Use Disorders
Brief Title: Telehealth Treatment for Opioid Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000034414; 1R61DA057675-01 (NIH)
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
Keywords: Harm Reduction; Medication for Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OUD Telehealth Platform (Experimental): Participants will be assigned to receive the OUD Telehealth Platform, which will be delivered remotely by research staff.
  Interventions: Behavioral: OUD Telehealth Platform

INTERVENTIONS:
Behavioral: OUD Telehealth Platform — The platform is intended to encourage engagement in treatment with medications for opioid use disorder (MOUD) through a chat dialogue with users

SUMMARY:
This study aims to use an Opioid Use Disorder (OUD) Telehealth Platform to reduce overdose events. This telehealth platform will be pilot tested to evaluate its preliminary efficacy in terms of motivating engagement in medications for OUD (MOUD), as well as its feasibility, acceptability and satisfaction to both first responders/providers and participants.

DETAILED DESCRIPTION:
The primary objective of the study is to assess effects of enrollment in a comprehensive telehealth platform, in adults with moderate or severe opioid use disorder with a history of at least one opioid overdose. Adults with moderate or severe opioid use disorder with a history of at least one opioid overdose will be enrolled and the primary endpoint will be attendance at first appointment for medication for opioid use disorder at 30 days.

Secondary aims include assessing engagement in the first MOUD appointment at 90 days and self-report of the number of subsequent overdose events at 30 and 90 days. Exploratory aims include feasibility of intervention, readiness and intention to engage in treatment, acceptability and satisfaction of intervention, and comparison of MOUD engagement with data from previous in-person studies.

ELIGIBILITY:
Inclusion Criteria:

* Can speak, read and write in English
* Provision of signed and dated informed consent form
* Have a history of at least one opioid overdose
* Screened positive for OUD, moderate or severe, based on the Diagnostic and Statistical Manual-5th Edition
* Have a working cell phone number and working device that can access a web browser and receive texts (i.e., smartphone, tablet or computer) OR be willing to use a device provided by the study team
* Can provide a working email address OR be willing to create one

Exclusion Criteria:

* Current use of buprenorphine, methadone, or naltrexone for a substance use disorder
* Pregnancy
* Known current suicide risk based on participant self-report
* On parole or incarcerated at time of enrollment based on participant self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Attendance for MOUD | Up to 30 Days
  Overall attendance will be measured by attendance (yes or no) at the first buprenorphine appointment within 30 days of referral.

SECONDARY OUTCOMES:
Engagement with MOUD | Up to 90 days
  Engagement will be measured by demonstrated maintained attendance with MOUD treatment within 90 days of referral.
Overdose Events at 30 Days | Up to 30 days
  A self-report of the number of subsequent overdose events at 30 days.
Overdose Events at 90 Days | Up to 90 days
  A self-report of the number of subsequent overdose events at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Heckmann, MD, MPH, MPA, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as part of the HEAL Initiative Consortium.
Time Frame: Following the close of the study and final reporting to funder.

REFERENCES:
- [Derived] Canty T, S Sabounchi N, Heimer R, Pantalon M, Ryus C, Buchanan L, Grewal M, Maffei J, D'Onofrio G, Heckmann R. Increasing timely access to evidence-based treatment for opioid use disorder using novel digital health and system dynamics modelling approaches: a study protocol. BMJ Open. 2025 Nov 4;15(11):e102796. doi: 10.1136/bmjopen-2025-102796. PMID 41193189